CLINICAL TRIAL: NCT01624038
Title: Phase 2 Study of Therapeutic Effect and Safety of Combined Hydroxyurea With Recombinant Human Erythropoietin.
Brief Title: Therapeutic Effect and Safety of Combined Hydroxyurea With Recombinant Human Erythropoietin.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohsen Saleh Elalfy, prof. Mohsen el alfy, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: huoepio
Record Dates: First submitted 2012-04-13; First posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Thalassemia Intermedia
Keywords: Hydroxyurea; Erythropoitin therapy; Thalassemia intermedia
MeSH Terms: conditions — beta-Thalassemia | interventions — Hydroxyurea; Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydroxyurea,blood transfusion (Active Comparator): Hydroxyurea (Myers-Squibb, USA) was administered in dosages ranging from 15 up to 35 mg/kg/day orally over 7 days/week.
  Interventions: Drug: hydroxyurea, blood transfusion
- Hydroxyurea, Epiao (Experimental): * Hydroxyurea (Myers-Squibb, USA) was administered in dosages ranging from 15 up to 35 mg/kg/day orally over 7 days/week. Hydroxyurea toxicity was defined as a white cell count of less than 2500/μL or a platelet count of less than 100,000/μL, in which case the drug was discontinued. White cell count and platelet count were determined on a monthly basis. Side effects such as nausea, vomiting, diarrhea, rashes, and malaise, experienced during the first 6 h after taking the HU will be considered as clinical toxicity.
  * Erythropiotien therapy (rHuEPO - Epiao) from 250 to 500 IU/kg rHuEPO subcutaneously three times a week.
  Interventions: Drug: Hydroxyurea ,Epiao

INTERVENTIONS:
Drug: Hydroxyurea ,Epiao — Hydroxyurea (Myers-Squibb, USA) was administered in dosages ranging from 15 up to 35 mg/kg/day orally over 7 days/week.
  Erythropiotien therapy (rHuEPO - Epiao) from 250 to 500 IU/kg rHuEPO subcutaneously three times a week.
  Arms: Hydroxyurea, Epiao
Drug: hydroxyurea, blood transfusion — * Hydroxyurea was administered in dosages ranging from 15 up to 35 mg/kg/day orally over 7 days/week. Hydroxyurea toxicity was defined as a white cell count of less than 2500/μL or a platelet count of less than 100,000/μL, in which case the drug was discontinued.
  Arms: Hydroxyurea,blood transfusion

SUMMARY:
The study hypothesis that treatment with Erythropoietin (EPO) combined with Human Erythropoietin (HUO) therapy will result in hematologic improvement in thalassemia intermedia patients.

Second is to determine whether any of the following correlate with improved hematologic response:

A decrease in hemolysis, as assayed by a decrease in LDH, compared to baseline levels,baseline Erythropoietin levels,baseline hemoglobin levels and baseline reticulocyte counts (or % circulating nucleated erythroblasts/100 WBCs).

Goal:

The aim is to assess the possibility of steady increase of hemoglobin levels in thalassemia intermedia patients by at least 1g/dl above baseline levels during therapy using Hydroxyurea and Erythropoietin, growth evaluation,quality of life (QoL) and decline transfusion requirements during study period. Also to report and compare adverse events with other published data regarding.

DETAILED DESCRIPTION:
To determine whether any of the following correlate with improved hematologic response:

A decrease in hemolysis, as assayed by a decrease in LDH, compared to baseline levels,baseline Erythropoietin levels,baseline hemoglobin level and baseline reticulocyte counts (or % circulating nucleated erythroblasts/100 WBCs).

To assess the possibility of steady increase of hemoglobin levels in thalassemia intermedia patients by at least 1g/dl above baseline levels during therapy using Hydroxyurea and Erythropoietin, growth evaluation , quality of life ( QoL ) and decline transfusion requirements during study period. Also to report and compare adverse events with other published data regarding.

THE following criteria are used when including the patient in the study:

Patients with thalassemia intermedia.Diagnosis based on genetic mutations, hemoglobin electrophoresis and characteristic clinical data at presentation. Patients requiring different transfusion requirements and not transfusion dependent.Patients having a baseline hemoglobin of less than or equal to 6-8g/dl.Patients with normal renal and liver function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thalassemia intermedia. Diagnosis based on genetic mutations, hemoglobin electrophoresis and characteristic clinical data at presentation.
* Require different transfusion requirements and not transfusion dependent.
* Have a baseline hemoglobin of less than or equal to 6-8g/dl.
* Patients with normal renal and liver function.

Exclusion Criteria:

* Evidence of active hepatitis (ALT > 5 times above ULN).
* Evidence of renal impairment (serum creatinine > ULN).
* Patients who are dependent on red blood cell transfusions.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Change in baseline transfusion frequency with increase of pre-transfusion hemoglobin | baseline and 6 month hemoglobin level and transfusion frequency
  Decrease in baseline transfusion frequency with increase of pre-transfusion hemoglobin by calculation of transfusion index and mean hemoglobin level

SECONDARY OUTCOMES:
Change in baseline quality of life assessment. | baseline and 6 month QOL questionaire
  Quality of life assessment using (QOL questionaire) at the begining and at 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen S Elalfy, professor, Principal Investigator — Ain Shams University
Locations (1):
- hematology clinic ,pediatrics hospital, Ain Shams University hospital, Cairo, Egypt

REFERENCES:
- [Derived] Elalfy MS, Adly AA, Ismail EA, Elhenawy YI, Elghamry IR. Therapeutic superiority and safety of combined hydroxyurea with recombinant human erythropoietin over hydroxyurea in young beta-thalassemia intermedia patients. Eur J Haematol. 2013 Dec;91(6):522-33. doi: 10.1111/ejh.12182. Epub 2013 Oct 5. PMID 23927461